CLINICAL TRIAL: NCT01720381
Title: Manual vs. Automated moNitoring Accuracy of GlucosE II (MANAGE II)
Brief Title: OptiScanner Versus Standard Blood Glucose Monitoring
Status: Completed | Type: Observational
Sponsor: OptiScan Biomedical Corporation (Industry)
Collaborators: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2001078
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Hyperglycemia
Keywords: monitoring; blood glucose; intensive care unit
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — One additional blood sample (4 ml)will be collected once a day, separated into Draw an additional ~ 4.0 mL from the subject into a syringe once per every 24 hour period. The study site will indicate where and at what time the sample was taken. This sample is placed into a sodium heparin tube, labeled with the subject number and sampling time and centrifuged on a refrigerated centrifuge. The gained plasma will be frozen at minus 70 degrees Celsius or less and may be used for potential analysis by the Sponsor, should an analysis of outliers indicate the potential presence of an interferent.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study is to demonstrate the accuracy of the OptiScanner in measuring blood glucose levels in critically ill patients when compared to a reference YSI 2300 STAT Plus and the Gem 3000, the reference standard for Erasme University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed consent.
* Age ≥ 18 years.
* Admitted to the ICU of Erasme University Hospital.
* Expected ICU stay of ≥ 3 days at the time of enrollment (as judged by the Principle Investigator).
* APACHE II score of ≥ 10, within the first 24 hours of ICU admission.
* Existing central venous catheter + arterial catheter.
* No participation in any other investigational interventional study while enrolled in this study.
* Hyperglycemia (BG > 150 mg/dl) at the time of admission.

Exclusion Criteria:

* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted to the intensive care unit (ICU) of Erasme University Hospital in Brussels, Belgium.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Glucose Prediction error | 1 year
  Percent (%) predicted error is the percent (%) error result of the OptiScanner on central venous blood from the superior cava versus the YSI and the GEM using arterial blood.

SECONDARY OUTCOMES:
Clarke Error Grid analysis | 1 year
  The Clarke Error Grid analysis shows the percentage of paired values falling within each zone between the glucose results of the OptiScanner on central venous versus the YSI and the GEM using arterial blood.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Preiser, MD, PhD, Principal Investigator — Erasme University Hospital
Locations (1):
- Erasme University Hospital, Brussels, Belgium

REFERENCES:
- [Derived] Righy Shinotsuka C, Brasseur A, Fagnoul D, So T, Vincent JL, Preiser JC. Manual versus Automated moNitoring Accuracy of GlucosE II (MANAGE II). Crit Care. 2016 Nov 25;20(1):380. doi: 10.1186/s13054-016-1547-3. PMID 27884157